CLINICAL TRIAL: NCT05807204
Title: Effect of a Multi-ingredient of L-Histidine, L-Serine, L-Carnosine and N-Acetylcysteine on Visceral Adiposity and Non-alcoholic Fatty Liver Disease in Individuals With Abdominal Obesity. Randomized, Parallel, Placebo Controlled, Triple Blind Study.
Brief Title: Effect of a Multi-ingredient on Visceral Adiposity and Non-alcoholic Fatty Liver Disease in Individuals With Abdominal Obesity
Acronym: FATHIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Centre de Diagnosi per la Imatge (Unknown); Laboratorio de Referencia Sud (Unknown); Centro OWLiver (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FATHIS
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Visceral Obesity; Non-Alcoholic Fatty Liver Disease
Keywords: Nutraceuticals; Visceral Obesity; NAFLD; Metabolic risk; L-histidine; L-serine; N-Acetylcysteine; L-carnosine; Glucose metabolism; Lipid metabolism; Hepatic steatosis; Hypertension
MeSH Terms: conditions — Obesity, Abdominal; Non-alcoholic Fatty Liver Disease; Fatty Liver; Hypertension | interventions — Serine; Carnosine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine (Experimental): Participants will daily consume the multi-ingredient (L-Histidine, L-Serine, L-Carnosine and N-Acetylcysteine) for 12 weeks.
  Interventions: Dietary Supplement: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine
- Placebo (Placebo Comparator): Participants will daily consume the placebo (maltodextrin) for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine
Dietary Supplement: Placebo — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Placebo

SUMMARY:
The aim of this study is to validate the efficacy of specific combination of different natural histidine-related amino acids in the reduction of visceral fat and liver steatosis, as well their associated comorbidities, in individuals with abdominal obesity.

DETAILED DESCRIPTION:
World Health Organization (WHO) defines obesity as an excess of fat accumulation in adipose tissues and in other metabolic organs, leading to serious health implications. Obesity is a rising issue whose prevalence has defined as a global pandemic or globesity (>30% world population) being responsible of millions of deaths annually. Also, obesity is related with several comorbidities such as non-alcoholic fatty liver disease (NAFLD), with a global prevalence of >25%. Thus, strategies to ameliorate obesity and NAFLD are critical to improve life expectancy and quality of life and to reduce the economic burden of both diseases.

Current therapies against obesity are mainly focused on weight loss, including lifestyle intervention, to modify eating behaviours and to promote physical activity. However, the compliance of patients with these therapies is small. In addition, there are some drugs to fight against these diseases. In obesity, these medical therapies are focused to decrease fat gastrointestinal absorption using lipase inhibitors with several side effects: faecal incontinence, abdominal cramping and raise in blood pressure. In NAFLD, medical therapies are designed to reduce insulin resistance, using pioglitazone and metformin. However, the European Medicines Agency (EMA) and the Food and Drug Administration (FDA) recommend avoiding pioglitazone use by its relationship with heart failure and cancer, and metformin provides just a modest improvement in NAFLD.

Thus, the finding of new and efficient therapeutic agents is highly desirable to combat these global diseases.

The main objective of this study is to evaluate the effect of daily intake of a specific combination of L-histidine, L-serine, L-carnosine and N-Acetylcysteine, in combination with dietary recommendations, on the amount of visceral fat in individuals with abdominal obesity.

The secondary objectives of this study are to evaluate the effect of daily intake of the multi-ingredient aforementioned in liver fat content and obesity related comorbidities.

Participants who fulfilled the inclusion and exclusion criteria will be randomly assigned to the intervention and control group.

During the study there will be 4 visits: a preselection visit (V0; day -7) and 3 study visits during the consumption of the treatments, which will take place on the first day of the study (V1; day 1 +/- 3 days; week 1), at 6 weeks of treatment (V2; day 44 +/- 3 day; week 6) and at 12 weeks of treatment (V3; day 90 +/- 3 days; week 12).

ELIGIBILITY:
Inclusion Criteria:

* Men older than 40 years.
* BMI ≥30.0 kg/m^2 and ≤35.0 kg/m^2
* Waist circumference ≥102 cm.
* Read, write and speak Catalan or Spanish.
* Sign the informed consent.

Exclusion Criteria:

* Present values of body mass index > 35 kg/m^2
* Present values of waist circumference > 150 cm.
* Present diabetes.
* Present dyslipidemia (LDL cholesterol ≥ 189 mg/dL and/or triglycerides ≥ 350 mg/dL).
* Present anemia.
* Taking supplements, multivitamin supplements or phytotherapeutic products that interfere with the treatment under study.
* Consume 4 or more Standard Beverage Units (SBU) daily or 28 SBU weekly.
* Be a smoker.
* Present any diagnosed liver disease other than NAFLD.
* Have lost more than 3 kg of weight in the last 3 months.
* Present food intolerances and/or allergies related to the study products, such as hypersensitivity to maltodextrin or N-Acetylcysteine.
* Presenting any chronic or autoimmune disease in clinical manifestation such as hepatitis, hyper or hypothyroidism or metabolic diseases.
* Follow a pharmacological treatment with immunosuppressants, cytotoxic agents, corticosteroids or other drugs that could cause hepatic steatosis or alter the measurements in the liver.
* Being participating or having participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.
* Follow a hypocaloric diet and/or pharmacological treatment for weight loss.
* Suffering from eating behavior disorders or psychiatric disorders.
* Being unable to follow study guidelines.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Change in Visceral Adiposity | Change from Baseline Visceral Adiposity at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Visceral fat content measured using a dual energy x-ray absorptiometry (DXA) scanner

SECONDARY OUTCOMES:
Change in Hepatic Steatosis | Change from Baseline Hepatic Steatosis at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Liver steatosis will be qualitative determined by ultrasound
Height (cm) | At Baseline
  Height measured with standardized method
Change in Weight (kg) | Change from Baseline Weight at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight measured with standardized method
Change in Body Mass Index (BMI) (Kg/m^2) | Change from Baseline Body Mass Index at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight and height will be combined to report BMI in kg/m^2
Change in Neck circumference (cm) | Change from Baseline Neck circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Neck circumference using a measuring tape
Change in Arm circumference (cm) | Change from Baseline Arm circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Arm circumference using a measuring tape
Change in Waist circumference (cm) | Change from Baseline Waist circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Waist circumference using a measuring tape
Change in Conicity Index | Change from Baseline Conicity Index at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight, height and waist circumference will be combined to report Conicity index.
Change in Systolic Blood Pressure (mm Hg) | Change from Baseline Systolic Blood Pressure at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Systolic blood pressure will be measured using an automatic sphygmomanometer
Change in Diastolic Blood Pressure (mm Hg) | Change from Baseline Systolic Blood Pressure at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Diastolic blood pressure will be measured using an automatic sphygmomanometer
Change in intestinal microbiota composition | Change from Baseline intestinal microbiota composition at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Metagenomic analysis in fecal samples. The bacteria DNA will be extracted and massive sequenced by the Ion Torrent platform.
Change of biomarkers of oxidative stress (8-OHdG, F2-isoprostanes) | Change from Baseline biomarkers of oxidative stress at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Biomarkers of oxidative stress will be evaluated in urine by standardized chemiluminescence methods
Change in serum glucose levels (mg/dL) | Change from Baseline serum glucose levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum glucose levels will be determined by standardized spectrophotometry methods
Change in serum total cholesterol (mg/dL) | Change from Baseline serum total cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Total cholesterol will be determined by standardized spectrophotometry methods
Change in serum high-density lipoprotein cholesterol (HDL-C,mg/dL) | Change from Baseline serum high-density lipoprotein cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  High-density lipoprotein cholesterol will be determined by standardized spectrophotometry methods
Change in serum low-density lipoprotein cholesterol (LDL-C, mg/dL) | Change from Baseline serum low-density lipoprotein cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Low-density lipoprotein cholesterol will be calculated using the Friedewald formula
Change in serum triglycerides (TG, mg/dL) | Change from Baseline serum triglycerides at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Triglycerides will be determined by standardized spectrophotometry methods
Change in serum alanine aminotransferase (ALT, U/L) | Change from Baseline serum alanine aminotransferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Alanine aminotransferase will be determined by standardized spectrophotometry methods
Change in serum aspartate aminotransferase (AST, U/L) | Change from Baseline serum aspartate aminotransferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Aspartate aminotransferase will be determined by standardized spectrophotometry methods
Change in serum gamma glutamyl transferase (GGT, U/L) | Change from Baseline serum gamma glutamyl transferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Gamma glutamyl transferase will be determined by standardized spectrophotometry methods
Change in serum insulin levels (mU/L) | Change from Baseline serum insulin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Insulin levels will be measured by standardized chemiluminescence methods.
Change in serum leptin levels (pg/mL) | Change from Baseline serum leptin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Leptin levels will be measured by standardized chemiluminescence methods
Change in serum adiponectin levels (ng/mL) | Change from Baseline serum adiponectin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Adiponectin levels will be measured by standardized chemiluminescence methods
Change in Adiponectin/Leptin ratio (numerical ratio) | Change from Baseline Adiponectin/Leptin ratio at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Adiponectin and leptin will be combined to report adiponectin/leptin ratio
Change in serum Monocyte chemoattractant protein-1 (MCP-1) levels (pg/mL) | Change from Baseline serum MCP-1 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  MCP-1 levels will be measured by standardized chemiluminescence methods
Change in plasma tumor necrosis factor alpha (TNF-alpha) levels (pg/mL) | Change from Baseline plasma TNF-alpha levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  TNF-alpha levels will be measured by standardized chemiluminescence methods
Change in plasma Interleukin 6 (IL-6) levels (pg/mL) | Change from Baseline plasma IL-6 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  IL-6 levels will be measured by standardized chemiluminescence methods
Change in plasma Interleukin 10 (IL-10) levels (pg/mL) | Change from Baseline plasma IL-10 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  IL-10 levels will be measured by standardized chemiluminescence methods
Change in plasma Intercellular Adhesion Molecule 1 (ICAM-1) levels (ng/mL) | Change from Baseline plasma ICAM-1 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  ICAM-1 levels will be measured by standardized chemiluminescence methods
Change in plasma Cluster of Differentiation 14 (CD14) levels (pg/mL) | Change from Baseline plasma CD14 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  CD14 levels will be measured by standardized chemiluminescence methods
Change in plasma oxidized low density lipoproteins (LDLox) levels (mU/L) | Change from Baseline plasma LDLox levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  LDLox levels will be measured by standardized chemiluminescence methods
Change in serum C-Reactive protein levels (mg/L) | Change from Baseline serum C-Reactive protein levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  C-Reactive protein levels will be determined by standardized spectrophotometry methods
Change in Histidine levels in blood (umol/L) | Change from Baseline Histidine levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum histidine levels will be determined by Liquid Chromatography coupled to tandem Mass Spectrometry
Change in Homeostatic Model Assessment from Insulin Resistance Index (HOMA-IR) | Change from Baseline HOMA-IR at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  HOMA-IR will be calculated using serum glucose and insulin levels.
Change in Fatty Liver Index (FLI) | Change from Baseline FLI at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  FLI will be calculated using BMI, waist circumference, serum triglycerides and gamma glutamyl transferase levels
Change in Triglyceride glucose index (TyG) | Change from Baseline TyG at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  TyG will be calculated using serum glucose and triglycerides levels
Change in Plasma atherogenic index | Change from Baseline Plasma atherogenic index at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Plasma atherogenic index will be calculated as the logarithm of the TG to HDL-c ratio
Change in Dietary habits | Change from Baseline Dietary habits at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Nutritional habits will be determined based on the results obtained from the 3-day dietary record.
Change in Physical activity | Change from Baseline Physical activity at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Physical activity will be evaluated through the International Physical Activity Questionnaire (IPAQ)-short for physical activity questionnaire
Change in concomitant medication | Change from Baseline concomitant medication at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  The consumption of concomitant medication by the volunteers will be controlled by the record of concomitant medication in the case report form
Change in the consumption of food supplements | Change from Baseline consumption of food supplements at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  The consumption of food supplements by the volunteers will be controlled by the record of food supplements in the case report form
Analysis of genetic polymorphisms | Single nucleotide polymorphisms (SNPs) in loci of genetic susceptibility to abdominal adiposity will be studied at 12 weeks after treatment for each of the two treatments (multi-ingredient and placebo)
  Single Nucleotide Polymorphisms (SNPs) in saliva samples will be analysed by Illumina sequencing
Change of Food Intake Biomarkers | Change from Baseline Food Intake Biomarkers at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Food Intake biomarkers will be evaluated in urine using Metabolomics analyses (UHPLC MS)
Adverse events | After 6 (V2) and 12 weeks (V3) of treatment period for each of the two treatments (multi-ingredient and placebo)
  Possible adverse events derived from taking study's products will be recorded in the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Escoté, PhD, Principal Investigator — Eurecat, Technology Centre of Catalonia
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus — http://eurecat.org